CLINICAL TRIAL: NCT06104059
Title: Ιntraoperative Administration of Opioids Guided by the Nociception Level Index NOL in Elective Laparoscopic Surgeries Under General Anesthesia: Effect on Opioid Consumption, Post-operative Pain and Patient Recovery
Brief Title: NOL Guided Analgesia During Elective Laparoscopic Surgery Under General Anesthesia
Acronym: NOLGADELS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Paraskevi Matsota, Prof of Anesthesiology, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NOLGADELS
Record Dates: First submitted 2023-10-22; First posted 2023-10-27 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Intraoperative Analgesia
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized clinical trial
Who Masked: Participant
Masking Description: Not aware of the study group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nociception level index (NOL™) (Active Comparator): The nociception level index NOL will be used in order to quide intraopertaive analgesia.
  Interventions: Device: Nociception level index (NOL™)
- Standard of care (Active Comparator): Intraoperative analgesia will be based on common practice, i.e. changes in hemodynamic parameters.
  Interventions: Other: Fentanyl

INTERVENTIONS:
Device: Nociception level index (NOL™) — If a NOL value >25 persists for >1 minute a bolus of iv fentanyl 0.5mcg/kg will be given and reassessment of the NOL value will continue every 5 minutes. If NOL index value: 10-25 is not reached within 10 minutes, fentanyl 0.5mcg/kg iv is re-administered.
  Arms: Nociception level index (NOL™)
Other: Fentanyl — Bolus doses of iv fentanyl 0.5 mcg/kg will be administered based on the judgment of the anesthesiologist in charge.
  Arms: Standard of care

SUMMARY:
The aim of this study is to investigate the hypothesis that the intraoperative use of the nociception level index NOL can reduce opioid consumption in adult patients undergoing elective laparoscopic surgeries under general anesthesia, as well as to explore its effect on post-operative pain and patient recovery.

DETAILED DESCRIPTION:
The study is a Prospective Randomized clinical trial. Adult patients (>18y) undergoing elective laparoscopic surgery under general anesthesia will be included.

The patients will be randomized using the "sealed envelope" randomization method into two groups.

Intervention group: in this group, the nociception level index NOL will be used in order to guide intraoperative analgesia. Control group: in this group standard anesthetic care will be provided. Analgesic demands will be treated with bolus doses of iv fentanyl.

All patients will receive the same general anesthesia induction regimen. Patients upon entering the operating room will have standard monitoring applied [Noninvasive Blood Pressure (NIBP), ECG, SpO2] and a venous line placed. The depth of anesthesia will also be monitored by using the BIS sensor and placement of the NOL sensor. Specifically, a sensor (Covidien, BIS™ monitoring system with 3.50 software) will be placed on the forehead (after cleaning with an rubbing alcohol solution) and an NOL sensor (Medasense Biometrics Ltd., PMD200™) on a finger on the opposite upper extremity to that on which the blood pressure cuff will beplaced. Neuromuscular blockade will also be monitored using a neurostimulator (Organon, TOF-Watch SX) to stimulate and record the response of the ulnar nerve to TOF. Before induction to general anesthesia, all patients receive an IV bolus 1mg of midazolam and preoxygenation is performed for 5 minutes with a mask (FiO2: 100%, FGF: 12 l/min). Induction to general anesthesia will be performed with propofol 2.5mg/kg iv and fentanyl 2mcg/kg iv and once a BIS <60 is achieved, rocuronium 0.6mg/kg iv will be administered. At the same time, the patient's ventilation is supported with a mask and bag (FiO2:100%). When TOF=0, endotracheal intubation will be performed. After intubation, maintenance of anesthesia will be achieved by administration of sevoflurane 0.7 MAC in 50% O2/Air and co-administration of iv propofol infusion (75-150mcg/kg/min) with target BIS: 40-60. Subsequently, 8 mg iv dexamethasone and 0.1 mg/kg iv morphine will be administered and an arterial catheter is placed for continuous blood pressure measurement. Before the surgical incision, fentanyl IV 1.5mcg/kg will be administered and the surgical incisions will be infiltrated with a 0.375% ropivacaine solution of 20ml. Intraoperatively, to achieve optimal analgesia, iv fentanyl will be administered according to the group to which the patient has been allocated, as described above. Half an hour before the end of the operation, 1g paracetamol iv and 4mg ondasetron iv will be administered and 20 minutes before the end of the surgical procedure, the propofol infusion will stop.

Reversal of peripheral neuromuscular blockade will be perfomed using sugammadex: 2-4mg/kg, depending on the indication of the neurostimulator. The patient will be extubated if TOF=4 & TOF ratio ≥0.9 and BIS >80. Subsequently, the patient will be transferred to the Post Anesthesia Care Unit (PACU).

In PACU, intensity of postoperative pain will be assessed every 15 minutes with the Visual analogue scale (VAS, 0-10) and for a score >4, morphine 1mg iv bolus will be administered (up to 0.15mg/kg morphine in total for each patient including the intraoperative dose) until the patient is released from PACU.

Patient recovery will be assessed using the Post Anesthesia Recovery Score (PAR-Score), i.e. the Modified Aldrete score initially as soon as the patient is transferred to the PACU and patients will be released from PACU once they have score ≥9. The length of stay in the PACU until a score ≥9 is reached will also be recorded.

Any events or adverse effects (respiratory depression, lethargy, nausea, vomiting, itching, etc.) will also be recorded in the PACU.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing planned laparoscopic surgery under general anesthesia.

Exclusion Criteria:

* Emergency surgery.
* Pregnancy.
* Drug or alcohol abuse in the last 6 months.
* Chronic opioid use or patients with chronic pain.
* Serious comorbidity [cardiac disease (atrial fibrillation, ventricular arrhythmias), liver or kidney disease]
* Obesity (BMI >35).
* Permanently implanted pacemaker.
* Patients with CNS disease.
* Allergy to any of the study drugs.
* Patients receiving anticholinergics agonists, α2-adrenergic agonists, β1-adrenergic antagonists, antiarrhythmic drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Intraoperative total consumption of opioids | Up to 30 minutes after the end of operation
  Intraoperative total consumption of opioids will be calculated in all patients.

SECONDARY OUTCOMES:
Postoperative administration of opioids in PACU | Until the patient is released from PACU (up to 24 hours)
  Total consumption of opioids will be calculated in all patients
Intensity of postoperative pain in PACU | Until the patient is released from PACU (up to 24 hours)
  In PACU, intensity of postoperative pain will be assessed every 15 minutes with the Visual analogue scale, a 10 points scale (0= no pain and 10= worst pain)

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of Anesthesiology, Attikon University Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No